CLINICAL TRIAL: NCT00061841
Title: Medical College of Georgia FitKid Project
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: FITKID (DK63391) (completed)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2010-01-13 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
MeSH Terms: interventions — Exercise

INTERVENTIONS:
Behavioral: exercise

SUMMARY:
This project will determine whether exposing youths to a "fitogenic" after-school environment that emphasizes vigorous exercise and healthy snacks will have a favorable effect on body composition (i.e., less fat tissue and more lean tissue), cardiovascular fitness and cardiovascular disease risk profile. The environmental intervention will be provided in nine schools in Augusta, Georgia, with another nine schools serving as non-intervention comparison schools. Children in the 3rd grade will be recruited to participate. They will be followed for 3 years, through the 5th grade. Measurements will be made at the beginning and end of each school year. The 2-hour after-school intervention will be offered every school day. It will consist of three components: (1) homework assistance; (2) a healthy snack; and (3) exercise designed to improve skills and fitness.

ELIGIBILITY:
3rd graders in schools chosen to participate.

Ages: 8 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 685 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Medical College of Georgia, Augusta, Georgia, United States

REFERENCES:
- [Derived] Yin Z, Moore JB, Johnson MH, Vernon MM, Gutin B. The impact of a 3-year after-school obesity prevention program in elementary school children. Child Obes. 2012 Feb;8(1):60-70. doi: 10.1089/chi.2011.0085. PMID 22799482